CLINICAL TRIAL: NCT04994509
Title: A Phase 3, Double-Blinded, Multicenter, Randomized Study to Evaluate Safety and Efficacy of Twice Yearly Long-Acting Subcutaneous Lenacapavir, and Daily Oral Emtricitabine/Tenofovir Alafenamide for Pre-Exposure Prophylaxis in Adolescent Girls and Young Women at Risk of HIV Infection
Brief Title: Pre-Exposure Prophylaxis Study of Lenacapavir and Emtricitabine/Tenofovir Alafenamide in Adolescent Girls and Young Women at Risk of HIV Infection
Acronym: PURPOSE 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GS-US-412-5624; DOH-27- 072021-6125 (Registry Identifier: South African National Clinical Trial Registry)
Record Dates: First submitted 2021-08-02; First posted 2021-08-06 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Pre-Exposure Prophylaxis of HIV Infection
MeSH Terms: interventions — lenacapavir; Injections, Subcutaneous; emtricitabine tenofovir alafenamide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Randomized Blinded Phase: Lenacapavir (Experimental): Participants will receive lenacapavir (LEN) 927 mg injection, every 26 weeks starting on Day 1 for up to approximately 52 weeks. Participants will also receive loading dose of LEN 600 mg, tablet, once daily on Day 1 and Day 2. Participants will receive placebo to match (PTM) emtricitabine/tenofovir disoproxil fumarate (F/TDF) or PTM emtricitabine/tenofovir alafenamide (F/TAF), once daily, up to approximately 52 weeks.
  Interventions: Drug: Oral Lenacapavir (LEN); Drug: Subcutaneous (SC) Lenacapavir (LEN); Drug: PTM F/TAF; Drug: PTM F/TDF
- Randomized Blinded Phase: F/TAF (Experimental): Participants will receive F/TAF, once daily up to approximately 52 weeks. Participants will also receive PTM LEN injection, every 26 weeks, starting on Day 1 up to approximately 52 weeks. Participants will receive PTM LEN tablet, once daily on Day 1 and Day 2.
  Interventions: Drug: F/TAF; Drug: Placebo SC LEN; Drug: PTM Oral LEN
- Randomized Blinded Phase: F/TDF (Experimental): Participants will receive F/TDF, once daily up to approximately 52 weeks. Participants will also receive PTM LEN injection, every 26 weeks starting on Day 1 up to approximately 52 weeks. Participants will receive PTM LEN tablet, once daily on Day 1 and Day 2.
  Interventions: Drug: F/TDF; Drug: Placebo SC LEN; Drug: PTM Oral LEN
- LEN Open-Label Extension (OLE) Phase (Experimental): After completion of the Blinded phase, participants will be offered entry into the LEN OLE Phase.
  Participants randomized to LEN will continue to receive LEN 927 mg injection, every 26 weeks until LEN becomes available or the sponsor elects to discontinue the study, whichever occurs first.
  Participants randomized to F/TAF or F/TDF will receive LEN 927 mg injection on OLE Day 1, Week 26, and every 26 weeks thereafter. Participants will also receive LEN 600 mg tablet on OLE Days 1 and 2.
  Interventions: Drug: Oral Lenacapavir (LEN); Drug: Subcutaneous (SC) Lenacapavir (LEN)
- Pharmacokinetic (PK) Tail Coverage Phase (Experimental): Participants who prematurely discontinue study drug in the randomized blinded phase will transition into the PK Tail Coverage phase.
  Participants will receive F/TDF, once daily, for 78 weeks beginning 26 weeks after the last LEN injection.
  Interventions: Drug: F/TDF

INTERVENTIONS:
Drug: Oral Lenacapavir (LEN) — Tablets administered orally without regard to food
  Other Names: GS-6207
  Arms: LEN Open-Label Extension (OLE) Phase; Randomized Blinded Phase: Lenacapavir
Drug: Subcutaneous (SC) Lenacapavir (LEN) — Administered via SC injections
  Other Names: GS-6207; Yeztugo®
  Arms: LEN Open-Label Extension (OLE) Phase; Randomized Blinded Phase: Lenacapavir
Drug: F/TAF — Tablets administered orally
  Other Names: Descovy®
  Arms: Randomized Blinded Phase: F/TAF
Drug: F/TDF — Tablets administered orally
  Other Names: Truvada®
  Arms: Pharmacokinetic (PK) Tail Coverage Phase; Randomized Blinded Phase: F/TDF
Drug: Placebo SC LEN — Administered via SC injections
  Arms: Randomized Blinded Phase: F/TAF; Randomized Blinded Phase: F/TDF
Drug: PTM Oral LEN — Tablets administered orally
  Arms: Randomized Blinded Phase: F/TAF; Randomized Blinded Phase: F/TDF
Drug: PTM F/TAF — Tablets administered orally
  Arms: Randomized Blinded Phase: Lenacapavir
Drug: PTM F/TDF — Tablets administered orally
  Arms: Randomized Blinded Phase: Lenacapavir

SUMMARY:
The goal of this study is to evaluate the efficacy of the study drugs, lenacapavir (LEN) and emtricitabine/tenofovir alafenamide (F/TAF) in preventing HIV infection, in adolescent girls and young women (AGYW).

The primary objective of this study is to evaluate the efficacy of LEN and F/TAF for HIV-1 PrEP in AGYW at risk of HIV-1 infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Incidence Phase

  * HIV-1 status unknown at initial screening and no prior human immunodeficiency virus (HIV)-1 testing within the last 3 months.
  * Sexually active (has had > 1 vaginal intercourse within the last 3 months) with cisgender male individuals (CGM).
* Randomized Phase

  * Negative fourth generation HIV-1 antibody (Ab)/antigen (Ag) test confirmed with central HIV-1 testing.
  * Estimated glomerular filtration rate (GFR) ≥ 60 mL/min at screening.
  * Body weight ≥ 35 kg.

Key Exclusion Criteria:

* Prior receipt of an HIV vaccine.
* Prior use of any long-acting systemic HIV pre-exposure prophylaxis (PrEP) or prior HIV postexposure prophylaxis (PEP) in the past 12 weeks.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender Female
Enrollment: 5368 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2028-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (28):
- South Africa (25):
  - Madibeng Centre for Research, Brits
  - Emavundleni Research Centre, Cape Town
  - Vuka Research Clinic, Cape Town
  - Desmond Tutu Health Foundation Clinical Trials Unit, Cape Town
  - Botha's Hill Clinical Research Site, HIV Prevention Research Unit, Durban
  - CAPRISA eThekwini Clinical Research Site, Durban
  - CAPRISA Vulindlela Clinical Research Site, Durban
  - MatCH Research Unit, Suite 1112, 11th Floor, Durban
  - Synergy Biomed Research Institute (SBRI), East London
  - Setshaba Research Centre, Gauteng
  - Wits Reproductive Health & HIV Institute (Wits RHI), Johannesburg
  - The Aurum Institute: Gavin J Churchyard Legacy Centre, Klerksdorp Clinical Research Centre, Klerksdorp
  - Perinatal HIV Research Unit (PHRU) Soweto Kliptown, Kliptown
  - Phoenix Clinical Research Site, South African Medical Research Council, HIV and Other Infectious Disease Research Unit, Kwa Zulu Natal
  - Verulam Clinical Research Site, South African Medical Research Council, HIV and Other Infectious Disease Research Unit, Kwa Zulu Natal
  - Tongaat Clinical Research Site, South African Medical Research Council, HIV and Other Infectious Disease Research Unit, Kwa Zulu Natal
  - Chatsworth Clinical Research Site, South African Medical Research Council, HIV and Other Infectious Disease Research Unit, Kwa Zulu Natal
  - Qhakaza Mbokodo Research Clinic, Ladysmith
  - Africa Health Research Institute, Mtubatuba
  - The Aurum Institute: Pretoria Clinical Research Centre, Pretoria
  - The Aurum Institute: Rustenburg Clinical Research Centre, Rustenburg
  - Desmond Tutu Health Foundation - Masiphumelele Research Office, Sunnydale
  - The Aurum Institute: Tembisa Clinical Research Centre, Tembisa
  - CAPRISA Umlazi Clinical Research Site, Umlazi
  - FPD-DTHF Ndevana Community Research Site, Vincent
- Uganda (3):
  - Makerere-Kalangala Clinical Research site, Kalangala
  - AMBSO Masaka Clinical Research site, Kyotera- Masaka Region
  - Makerere University- John Hopkins University (MU-JHU) Mityana Research Site (MU-JHU) Care Ltd, Mityana Town

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bekker LG, Das M, Abdool Karim Q, Ahmed K, Batting J, Brumskine W, Gill K, Harkoo I, Jaggernath M, Kigozi G, Kiwanuka N, Kotze P, Lebina L, Louw CE, Malahleha M, Manentsa M, Mansoor LE, Moodley D, Naicker V, Naidoo L, Naidoo M, Nair G, Ndlovu N, Palanee-Phillips T, Panchia R, Pillay S, Potloane D, Selepe P, Singh N, Singh Y, Spooner E, Ward AM, Zwane Z, Ebrahimi R, Zhao Y, Kintu A, Deaton C, Carter CC, Baeten JM, Matovu Kiweewa F; PURPOSE 1 Study Team. Twice-Yearly Lenacapavir or Daily F/TAF for HIV Prevention in Cisgender Women. N Engl J Med. 2024 Oct 3;391(13):1179-1192. doi: 10.1056/NEJMoa2407001. Epub 2024 Jul 24. PMID 39046157
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-412-5624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8402 participants were screened. Out of 8402, 8094 participants had at least 1 non-missing HIV-1 diagnosis based on HIV test results from a central laboratory. Therefore, 8094 participants were considered for screening in the Incidence Phase and were included in the All Screened Set.
Pre-assignment Details: Participants were enrolled at study sites in South Africa and Uganda. Data submitted represent primary analysis performed on data collected by the Primary Analysis Completion Date (Per pre-specified analysis, this is the date by when at least 50% of the planned randomized participants were followed up for at least 52 weeks in the study or prematurely discontinued from the study). Complete data will be submitted within 1 year of actual study completion date.
Groups:
- Randomized Blinded Phase: Lenacapavir: Participants received lenacapavir (LEN) 927 mg subcutaneous (SC) injection, every 26 weeks, starting on Day 1 up to approximately 52 weeks. Participants also received loading dose of LEN 600 mg tablet orally, once daily on Day 1 and Day 2. Participants received placebo to match (PTM) emtricitabine/tenofovir disoproxil fumarate (F/TDF) tablet or PTM emtricitabine/tenofovir alafenamide (F/TAF) tablet orally, once daily, up to approximately 52 weeks.
- Randomized Blinded Phase: F/TAF: Participants received F/TAF tablet on Day 1 orally, once daily up to approximately 52 weeks. Participants also received PTM LEN SC injection every 26 weeks starting on Day 1 up to approximately 52 weeks and PTM LEN tablet, orally, once daily on Day 1 and Day 2.
- Randomized Blinded Phase: F/TDF: Participants received F/TDF tablet on Day 1 orally, once daily up to approximately 52 weeks. Participants also received PTM LEN SC injection, every 26 weeks, starting on Day 1 up to approximately 52 weeks and PTM LEN tablet, orally, once daily on Day 1 and Day 2.
Period: Overall Study
Arm/Group | Randomized Blinded Phase: Lenacapavir | Randomized Blinded Phase: F/TAF | Randomized Blinded Phase: F/TDF
Started | 2150 | 2145 | 1073
Completed (Completed = Discontinued and entered into Open-label F/TDF Treatment Phase.) | 94 | 77 | 37
Not Completed | 2056 | 2068 | 1036
Not completed — Still on Study (Participants Continuing in Randomized Blinded Phase) | 1909 | 1910 | 937
Not completed — Withdrew Consent | 73 | 72 | 46
Not completed — Lost to Follow-up | 39 | 36 | 26
Not completed — HIV-1 Infection | 4 | 20 | 12
Not completed — Investigator's Discretion | 9 | 8 | 11
Not completed — Randomized but Never Treated | 10 | 10 | 3
Not completed — Pregnancy | 5 | 5 | 0
Not completed — Death | 0 | 5 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Non-compliance With Study Drug | 1 | 1 | 1
Not completed — Withdrew Assent | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized Blinded Phase Safety Analysis Set included all participants who received at least 1 dose of any study drug.
Groups:
- Randomized Blinded Phase: Lenacapavir: Participants received LEN 927 mg SC injection, every 26 weeks starting on Day 1 up to approximately 52 weeks. Participants also received loading dose of LEN 600 mg tablet orally, once daily on Day 1 and Day 2. Participants received PTM F/TDF tablet or PTM F/TAF tablet orally, once daily, up to approximately 52 weeks.
- Randomized Blinded Phase: F/TAF: Participants received F/TAF tablet on Day 1 orally, once daily up to approximately 52 weeks. Participants also received PTM LEN SC injection every 26 weeks starting on Day 1 up to approximately 52 weeks and PTM LEN tablet orally once daily on Day 1 and Day 2.
- Randomized Blinded Phase: F/TDF: Participants received F/TDF tablet on Day 1 orally, once daily up to approximately 52 weeks. Participants received PTM LEN SC injection, every 26 weeks starting on Day 1 up to approximately 52 weeks and PTM LEN tablet orally once daily on Day 1 and Day 2.
- Total: Total of all reporting groups
Arm/Group | Randomized Blinded Phase: Lenacapavir | Randomized Blinded Phase: F/TAF | Randomized Blinded Phase: F/TDF | Total
Number analyzed (Participants) | 2140 | 2135 | 1070 | 5345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 287 | 256 | 125 | 668
  Between 18 and 65 years | 1853 | 1879 | 945 | 4677
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2.2) | 21 (2.1) | 21 (2.1) | 21 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2140 | 2135 | 1070 | 5345
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2140 | 2135 | 1070 | 5345
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2137 | 2134 | 1068 | 5339
  White | 0 | 0 | 0 | 0
  More than one race | 3 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 1811 | 1788 | 909 | 4508
  Uganda | 329 | 347 | 161 | 837

OUTCOME MEASURES:

1. Primary Outcome: Incidence Phase: Recent Infection Testing Algorithm (RITA) Estimate of the Background Human Immunodeficiency-1 Virus Infection Incidence Rate (bHIV) Per 100 Person Years (PY)
Description: bHIV per 100 PY in the Incidence Phase was calculated using RITA.
  The RITA incorporated HIV-1 testing results and recency assay testing results to estimate the bHIV. Recency assay testing was performed for participants in the All Screened Set found to have HIV-1 infection at the Incidence Phase Screening Visit as defined below. Participants were considered to have recent HIV-1 infection if the normalized optical density (ODn) was below 1.5 threshold using the Sedia limiting antigen avidity enzyme immunoassay (LAg-EIA) and the HIV-1 RNA (viral load) was > 75 copies/mL of blood.
  HIV-1 infection was defined as participants having at least one of the following central lab results at the Incidence Phase screening visit:
  * Positive HIV-1/2 differentiation Ab, OR
  * Positive HIV-1 ribonucleic acid (RNA) qualitative test, OR
  * HIV-1 RNA quantitative test ≥200 copies/mL.
Time Frame: Incidence Phase Screening Visit (Day 1)
Population: Participants in the All Screened Set were analyzed. The All Screened Set included all participants who were screened for HIV-1 in the Incidence Phase and had a non-missing HIV-1 diagnosis based on HIV test results at Incidence Phase screening. As the outcome measure was assessed prior to Randomized Blinded Phase, the data is reported in one arm consisting of all participants screened in Incidence Phase.
Measure: Number (95% Confidence Interval); unit: HIV-1 events per 100 person-years
Groups:
- Participants Screened for HIV-1 in Incidence Phase: Participants screened for HIV-1 infection and having a non-missing HIV-1 diagnosis based on results of HIV testing conducted at Incidence Phase screening.
Arm/Group | Participants Screened for HIV-1 in Incidence Phase
Number analyzed (Participants) | 8094
HIV-1 events per 100 person-years | 2.407 [1.815 to 3.191]

2. Primary Outcome: Randomized Blinded Phase: HIV-1 Incidence Reported Per 100 PY for LEN and F/TAF Compared to Participants in All Screened Set
Description: HIV-1 incidence per 100 PY for LEN and F/TAF was calculated as the number of participants who acquired HIV-1 divided by the total of a) for participants not diagnosed with HIV-1, sum of all duration of follow-up time in years, while at risk of HIV-1 infection (where a year is 365.25 days) and b) for participants diagnosed with HIV-1, sum of all duration of follow-up time up to confirmed HIV-1 diagnoses.
  HIV-1 diagnosis was determined by an HIV adjudication committee who reviewed potential HIV-1 infection events in the randomized participants. The committee, in a blinded, consistent, and unbiased manner, determined whether HIV test results confirmed HIV-1 infection and determined the date of diagnosis for each case, defined as the date of the earliest study visit with evidence of HIV infection considering both prospective HIV testing and back-testing of archived samples.
  bHIV incidence per 100 PY in All Screened Set was estimated as described in outcome measure#1.
Time Frame: When at least 50% of the participants completed 52 weeks of follow-up after randomization or permanently discontinued from the study (maximum 143 weeks)
Population: Participants in the LEN and F/TAF groups in the Full Analysis Set (FAS) were analyzed. The FAS included all randomized participants who received at least 1 dose of any study drug and had not been diagnosed with HIV-1 on or prior to the first dose date. Per prespecified analysis, HIV-1 incidence for this outcome measure was reported only for participants who received LEN and F/TAF. The HIV-1 incidence was compared with participants in All Screened Set.
Measure: Number (95% Confidence Interval); unit: HIV-1 events per 100 person-years
Groups:
- Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis: Participants screened for HIV-1 infection and having a non-missing HIV-1 diagnosis based on HIV test results at Incidence Phase screening.
Arm/Group | Randomized Blinded Phase: Lenacapavir | Randomized Blinded Phase: F/TAF | Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis
Number analyzed (Participants) | 2134 | 2136 | 8094
HIV-1 events per 100 person-years | 0.000 [0.000 to 0.190] | 2.018 [1.435 to 2.759] | 2.407 [1.815 to 3.191]
Statistical Analysis 1: Comparison: Randomized Blinded Phase: Lenacapavir vs Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis; Null Hypothesis 01: LEN/bHIV>= 1; Null hypothesis was to be rejected if HIV-1 incidence in LEN was significantly lower than bHIV; Test type: Superiority; p < 0.0001, Likelihood ratio test — p-value for rate ratio vs bHIV is from likelihood ratio test; Rate Ratio = 0.000, 95% CI 2-sided [0.000 to 0.042] — Confidence Interval (CI) for rate ratio vs bHIV is from a likelihood-based method
Statistical Analysis 2: Comparison: Randomized Blinded Phase: Lenacapavir vs Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis; Null Hypothesis 02: LEN/bHIV>= 0.8; Null hypothesis was to be rejected if HIV-1 incidence in LEN was significantly and at least 20% lower than bHIV; Test type: Superiority; p < 0.0001, Likelihood ratio test — p-value for rate ratio vs bHIV is from likelihood ratio test; Rate Ratio = 0.000, 95% CI 2-sided [0.000 to 0.042] — CI for rate ratio vs bHIV is based on a likelihood-based method
Statistical Analysis 3: Comparison: Randomized Blinded Phase: F/TAF vs Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis; Null Hypothesis 03: F/TAF/bHIV>= 1; Null hypothesis was to be rejected if HIV-1 incidence in F/TAF was significantly lower than bHIV; Test type: Superiority; p = 0.20697, Wald test — p-value for rate ratio vs bHIV is from Wald test; Rate Ratio = 0.839, 95% CI 2-sided [0.550 to 1.279] — CI for rate ratio vs bHIV is based on the delta method
Statistical Analysis 4: Comparison: Randomized Blinded Phase: F/TAF vs Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis; Null Hypothesis 04: F/TAF/bHIV>= 0.8; Null hypothesis was to be rejected if HIV-1 incidence in F/TAF was significantly and at least 20% lower than bHIV; Test type: Superiority; p = 0.58674, Wald test — p-value for rate ratio vs bHIV is from Wald test; Rate Ratio = 0.839, 95% CI 2-sided [0.550 to 1.279] — CI for rate ratio vs bHIV is based on the delta method

3. Secondary Outcome: Randomized Blinded Phase: HIV-1 Incidence Reported Per 100 PY for LEN, F/TAF and F/TDF
Description: HIV-1 incidence per 100 PY was calculated as the number of participants who acquired HIV-1 divided by the total of a) for participants not diagnosed with HIV-1, sum of all duration of follow-up time in years, while at risk of HIV-1 infection (where a year is 365.25 days) and b) for participants diagnosed with HIV-1, sum of all duration of follow-up time up to confirmed HIV-1 diagnoses.
  HIV-1 diagnosis was determined by an HIV adjudication committee who reviewed potential HIV-1 infection events in the randomized participants. The committee, in a blinded, consistent, and unbiased manner, determined whether HIV test results confirmed HIV-1 infection and determined the date of diagnosis for each case, defined as the date of the earliest study visit with evidence of HIV infection considering both prospective HIV testing and back-testing of archived samples.
Time Frame: as for outcome 2
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: HIV-1 events per 100 person-years
Arm/Group | Randomized Blinded Phase: Lenacapavir | Randomized Blinded Phase: F/TAF | Randomized Blinded Phase: F/TDF
Number analyzed (Participants) | 2134 | 2136 | 1068
HIV-1 events per 100 person-years | 0.000 [0.000 to 0.190] | 2.018 [1.435 to 2.759] | 1.685 [0.963 to 2.737]
Statistical Analysis 1: Comparison: Randomized Blinded Phase: Lenacapavir vs Randomized Blinded Phase: F/TDF; Test type: Superiority; p < 0.0001, Poisson model — p-value for rate ratio vs F/TDF is from an exact conditional Poisson model; Rate Ratio = 0.000, 95% CI 2-sided [0.000 to 0.101] — CI is from an exact conditional Poisson model
Statistical Analysis 2: Comparison: Randomized Blinded Phase: F/TAF vs Randomized Blinded Phase: F/TDF; Test type: Superiority; p = 0.72820, Poisson model — p-value for rate ratio vs F/TDF is from a Poisson model; Rate Ratio = 1.198, 95% CI 2-sided [0.669 to 2.143] — CI is from a Poisson model
Statistical Analysis 3: Comparison: Randomized Blinded Phase: Lenacapavir vs Randomized Blinded Phase: F/TDF; Test type: Other — Comparability to F/TDF is defined as the HIV-1 incidence in the LEN group at most 0.8/100 PY higher than in the F/TDF group; p < 0.0001, Hybrid approach — p-value for rate difference vs F/TDF is based on a hybrid approach; Rate Difference = -1.685, 95% CI 2-sided [-2.737 to -0.939] — Exact CI is based on a hybrid approach
Statistical Analysis 4: Comparison: Randomized Blinded Phase: F/TAF vs Randomized Blinded Phase: F/TDF; Test type: Other — Comparability to F/TDF is defined as the HIV-1 incidence in the F/TAF group at most 0.8/100 PY higher than in the F/TDF group; p = 0.20900, Hybrid approach — p-value for rate difference vs F/TDF is based on a hybrid approach; Rate Difference = 0.333, 95% CI 2-sided [-0.869 to 1.367] — Exact CI is based on a hybrid approach

4. Secondary Outcome: Randomized Blinded Phase: HIV-1 Incidence Among Participants Adherent to LEN
Description: A participant was defined as adherent to LEN if they have received all per-protocol administrations of LEN within 28 weeks since the previous administration. The incidence of HIV-1 infection per 100 PY calculation is defined in outcome measure #2.
Time Frame: as for outcome 2
Population: Participants in the Full Analysis Set who were adherent to LEN were analyzed.
Measure: Number (95% Confidence Interval); unit: HIV-1 events per 100 person-years
Groups:
- Randomized Blinded Phase: Lenacapavir: Participants received LEN 927 mg SC injection every 26 weeks starting on Day 1 up to approximately 52 weeks. Participants also received loading dose of LEN 600 mg tablet orally, once daily on Day 1 and Day 2. Participants received PTM F/TDF tablet or PTM F/TAF tablet orally, once daily, up to approximately 52 weeks.
Arm/Group | Randomized Blinded Phase: Lenacapavir
Number analyzed (Participants) | 1973
HIV-1 events per 100 person-years | 0.000 [0.000 to 0.214]

5. Secondary Outcome: Randomized Blinded Phase: Percentage of Participants Adherent to F/TAF in HIV-1 Diagnosed Participants and Their Matched Controls
Description: A participant's adherence to F/TAF was measured by tenofovir diphosphate (TFV-DP) in dried blood spot (DBS) samples, where <450 fmol/punch associates with an adherence of <2 days per week. The data is reported in two categories: low adherence (<2 days per week) and not low adherence (>= 2 days per week).
Time Frame: as for outcome 2
Population: The dried blood spot (DBS) Case-Control Analysis Set included all randomized participants who took at least 1 dose of study drug, were diagnosed with HIV-1 or were selected as a matched control (with no diagnosis of HIV-1) for a participant with HIV-1 and have at least 1 non-missing DBS concentration value reported by the DBS laboratory.
  Per pre-specified analysis, the data is reported in a subset of participants in the F/TAF arm with and without HIV-1 diagnosis.
Measure: Number; unit: percentage of participants
Groups:
- Randomized Blinded Phase: F/TAF (Participants With HIV-1 Diagnosis): Participants who were diagnosed with HIV-1 received F/TAF tablet on Day 1 orally, once daily up to approximately 52 weeks. Participants also received PTM LEN SC injection every 26 weeks starting on Day 1 up to approximately 52 weeks and PTM LEN tablet orally once daily on Day 1 and Day 2.
- Randomized Blinded Phase: F/TAF (Matched Controls - Participants With No HIV-1 Diagnosis): Participants who were selected as matched controls to participants with HIV-1, but did not have HIV-1 diagnosis. Participants received F/TAF tablet on Day 1 orally, once daily up to approximately 52 weeks. Participants also received PTM LEN SC injection every 26 weeks starting on Day 1 up to approximately 52 weeks and PTM LEN tablet orally once daily on Day 1 and Day 2.
Arm/Group | Randomized Blinded Phase: F/TAF (Participants With HIV-1 Diagnosis) | Randomized Blinded Phase: F/TAF (Matched Controls - Participants With No HIV-1 Diagnosis)
Number analyzed (Participants) | 37 | 159
percentage of participants
  Low (< 2 days/Week) | 91.9 | 65.9
  Not Low (>= 2 days/Week) | 8.1 | 34.1
Statistical Analysis 1: Comparison: Randomized Blinded Phase: F/TAF (Participants With HIV-1 Diagnosis) vs Randomized Blinded Phase: F/TAF (Matched Controls - Participants With No HIV-1 Diagnosis); Test type: Superiority; p = 0.0006, ExactConditionalLogisticRegressionModel — p-value is from exact conditional logistic regression model; Exact Odds Ratio = 9.00, 95% CI 2-sided [2.06 to 83.36] — Exact odds ratio and and CI are from exact conditional logistic regression model

6. Secondary Outcome: Randomized Blinded Phase: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as 1 or both of the following:
  * Any adverse events (AEs) leading to premature discontinuation of study drug, or
  * Any AEs with an onset date on or after the study drug start date and no later than the last exposure date after permanent discontinuation of the study drug.
  An AE was any untoward medical occurrence in a clinical study participant administered a study drug that did not necessarily had a causal relationship with the treatment.
Time Frame: When all participants have a minimum of 52 weeks of exposure to study drug or permanent discontinuation, whichever occurs first (maximum approximately 3 years)
Reporting Status: Not Posted

7. Secondary Outcome: Randomized Blinded Phase: Percentage of Participants Experiencing Clinically Significant Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any post-baseline visit, up to and including the last exposure date for participants who permanently discontinued study drug, or the last available date in the database snapshot for participants who were still on treatment at the time of an analysis.
Time Frame: as for outcome 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events: When at least 50% of the participants completed 52 weeks of follow-up after randomization or permanently discontinued from the study (maximum 143 weeks)
Description: All-cause Mortality: The All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse Events: The Randomized Blinded Phase Safety Analysis Set included all participants who received at least 1 dose of any study drug.
Groups:
- Randomized Blinded Phase: Lenacapavir: Participants received LEN 927 mg SC injection, every 26 weeks starting on Day 1 up to approximately 52 weeks. Participants also received loading dose of LEN 600 mg tablet orally, once daily on Day 1 and Day 2. Participants also received PTM F/TDF tablet or PTM F/TAF tablet orally, once daily, up to approximately 52 weeks.
- Randomized Blinded Phase: F/TDF: Participants received F/TDF tablet on Day 1 orally, once daily up to approximately 52 weeks. Participants also received PTM LEN SC injection, every 26 weeks starting on Day 1 up to approximately 52 weeks and PTM LEN tablet orally once daily on Day 1 and Day 2.
Arm/Group | Randomized Blinded Phase: Lenacapavir | Randomized Blinded Phase: F/TAF | Randomized Blinded Phase: F/TDF
All-Cause Mortality (participants affected / at risk) | 0/2150 | 6/2145 | 0/1073
Serious Adverse Events (participants affected / at risk) | 59/2140 | 85/2135 | 35/1070
Other Adverse Events (participants affected / at risk) | 1757/2140 | 1550/2135 | 756/1070
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Blinded Phase: Lenacapavir (N=2140) | Randomized Blinded Phase: F/TAF (N=2135) | Randomized Blinded Phase: F/TDF (N=1070)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1
Brain empyema (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 1
Injection site abscess (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Malaria (Infections and infestations) | 3 | 5 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 3 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 2 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2 | 2 | 0
Abortion of ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 15 | 28 | 9
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 3 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 1
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Device dislocation (Product Issues) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 2 | 4 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 2 | 3 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Threatened uterine rupture (Reproductive system and breast disorders) | 0 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Victim of homicide (Social circumstances) | 0 | 2 | 0
Victim of sexual abuse (Social circumstances) | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Blinded Phase: Lenacapavir (N=2140) | Randomized Blinded Phase: F/TAF (N=2135) | Randomized Blinded Phase: F/TDF (N=1070)
Diarrhoea (Gastrointestinal disorders) | 133 | 161 | 67
Nausea (Gastrointestinal disorders) | 144 | 234 | 142
Vomiting (Gastrointestinal disorders) | 125 | 235 | 107
Injection site nodule (General disorders) | 1365 | 347 | 183
Injection site pain (General disorders) | 669 | 521 | 237
Injection site swelling (General disorders) | 96 | 121 | 50
Genitourinary chlamydia infection (Infections and infestations) | 300 | 317 | 129
Genitourinary tract gonococcal infection (Infections and infestations) | 141 | 157 | 66
Upper respiratory tract infection (Infections and infestations) | 271 | 274 | 121
Urinary tract infection (Infections and infestations) | 307 | 304 | 163
Vulvovaginal candidiasis (Infections and infestations) | 146 | 172 | 67
Dizziness (Nervous system disorders) | 120 | 141 | 79
Headache (Nervous system disorders) | 285 | 351 | 155
Vaginal discharge (Reproductive system and breast disorders) | 166 | 191 | 87

LIMITATIONS AND CAVEATS:
Due to data monitoring committee recommendation to stop the study early if the prespecified evaluation criteria were met, this is the date by when at least 50% of the participants were followed up for at least 52 weeks in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04994509/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04994509/SAP_001.pdf